CLINICAL TRIAL: NCT06635408
Title: Cystatin c as a Predictive Biomarker of Acute Kidney Injury and Neurological Outcomes in Aneurysmal Subarachnoid Haemorrhage Patients
Brief Title: Cystatin c: a Biomarker of AKI in Aneurysmal Subarachnoid Haemorrhage Patients
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Ayman, principle investigator, Alexandria University
Other Study IDs: 9222704
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Delayed cerebral ischemia; Angiographic vasospasm; Aneurysmal subarachnoid hemorrhage
MeSH Terms: conditions — Acute Kidney Injury; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aki group: Cystatin c biomarker will be assessed to predict occurrence of early acute kidney injury
  Interventions: Diagnostic Test: cystatin c
- Non-Aki group: participants in this group will not develop acute kidney injury throughout the study duration
  Interventions: Diagnostic Test: cystatin c

INTERVENTIONS:
Diagnostic Test: cystatin c — a biomarker to assess renal function

SUMMARY:
The goal of this observational study is to assess cystatin c as a predictive biomarker of early acute kidney injury in aneurysmal subarachnoid hemorrhage patients. The main question it aims to answer is:

- Does cystatin c biomarker can predict early acute kidney injury in aneurysmal subarachnoid hemorrhage patients?

Participants will be grouped into Aki and Non-Aki groups based on RIFLE criteria and Cystatin c biomarker will be tested to answer the study question.

ELIGIBILITY:
Inclusion Criteria:

* Patient admission to hospital within 48 hours of subarachnoid haemorrhage onset.
* Subarachnoid haemorrhage caused by intracranial aneurysm rupture and is confirmed via computed tomography angiography (CTA).
* Medical treatment, microsurgical clipping, or interventional endovascular treatment of aneurysm is performed within 48 hours of subarachnoid haemorrhage onset.

Exclusion Criteria:

* Prior onset of subarachnoid haemorrhage or other neurological diseases such as ischemic stroke, hemorrhagic stroke, or severe head trauma.
* Systemic diseases, such as chronic liver diseases, chronic lung diseases, chronic heart failure, thyroid diseases and cancer.
* Renal impairment at time of admission (creatinine-based eGFR less than 60 ml/min per 1.73 m2 body surface area).
* Patients who are hemodynamically unstable at time of admission.
* Mortality within 10 days after admission (duration of study).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Aneurysmal subarachnoid hemorrhage patients
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 6 days
  stages "risk" and "injury" are considered early AKI

SECONDARY OUTCOMES:
Adverse neurological outcomes | 10 days all except mortality within 28 days
  Delayed cerebral ischemia Angiographic vasospasm Hydrocephalus Infection Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A El Erian, Professor, Study Chair — Alexandria University; Ashraf A Abdelhalim, Professor, Study Chair — Alexandria University; Sherif M El Hadi, Professor, Study Chair — Alexandria University
Locations (1):
- Faculty of medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
I keep the IPD information of study participants, based on principle of confidentiality Disclosure after participant permission is allowed

REFERENCES:
- [Background] Wang RR, He M, Gui X, Kang Y. A nomogram based on serum cystatin C for predicting acute kidney injury in patients with traumatic brain injury. Ren Fail. 2021 Dec;43(1):206-215. doi: 10.1080/0886022X.2021.1871919. PMID 33478333
- See also: An nih link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7833079/